CLINICAL TRIAL: NCT06243471
Title: "Hallux Abductus Valgus and Extensor Hallux Longus: Relationship Between Them, Preoperative and Postoperative Assessment, Pressure Platform and Treatment by MIS Surgery"
Brief Title: Hallux Abductus Valgus and Extensor Hallux Longus; Treatment by MIS Surgery
Acronym: HAV-EHL-MIS
Status: Completed | Type: Observational
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Other Study IDs: UCV/2022-2023/035
Record Dates: First submitted 2024-01-19; First posted 2024-02-06 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-07

CONDITIONS: Hallux Valgus and Bunion
Keywords: minimal incision surgery; Tenotomy; Extensor hallucis longus; Hallux Abducts Valgus
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Minimally Invasive Surgery Group with Zigzag EHL Tenotomy
  Interventions: Procedure: Minimally invasive procedures for the Hallux Abductus Valgus and a zig-zag tenotomy for the extensus hallux longus.
- Group 2: Minimally Invasive Surgery Group without Zig-zag EHL Tenotomy
  Interventions: Procedure: Minimally invasive procedures for the Hallux Abductus Valgus.

INTERVENTIONS:
Procedure: Minimally invasive procedures for the Hallux Abductus Valgus. — Minimally invasive procedures for the Hallux Abductus Valgus
  Groups: Group 2
Procedure: Minimally invasive procedures for the Hallux Abductus Valgus and a zig-zag tenotomy for the extensus hallux longus. — Minimally invasive procedures for the Hallux Abductus Valgus and a zig-zag tenotomy for the extensus hallux longus.
  Groups: Group 1

SUMMARY:
The goal of this clinical trial is to investigate the relationship between Hallux Abductus Valgus (HAV) and the hyperextension of the Extensor Hallucis Longus (EHL) tendon. The study aims to understand the efficacy of MIS surgery in treating foot deformities like HAV and to evaluate the impact of EHL tendon hyperextension on this condition.

The main questions this study aims to answer are:

* How does the hyperextension of the EHL tendon correlate with the presence and severity of HAV?
* What is the effectiveness of MIS surgery in correcting HAV deformities and addressing issues related to EHL tendon hyperextension? Participants in this study will undergo pre-surgical evaluation to assess the severity of HAV and measure the extent of EHL tendon hyperextension using pressure platform analysis and other relevant clinical measures. During the MIS surgery, participants will receive treatment targeted at correcting HAV, possibly involving partial tenotomy.

If there is a comparison group: Researchers will compare individuals who undergo MIS surgery for HAV correction with a control group not receiving this intervention. The comparison aims to assess the effects of MIS surgery on both HAV correction and the relationship between EHL tendon hyperextension and the deformity.

This study endeavors to shed light on the relationship between HAV and EHL tendon hyperextension, the effectiveness of MIS surgery in addressing these issues, and potentially pave the way for improved surgical techniques in treating foot pathologies.

DETAILED DESCRIPTION:
Main Objective: To analyze the effectiveness of incomplete zig-zag tenotomy of the EHL combined with minimally invasive foot surgery for the correction of moderate and severe hallux abducts valgus (HAV).

Secondary Objectives:

Compare pre-surgical and post-surgical plantar pressure changes. Determine American Orthopaedic Foot & Ankle Society Scale (AOFAS scale) values pre-surgery and post-surgery.

Compare the improvement in post-surgical results of angles: HAV, Intermetatarsal Angle (AIM),Proximal Articular Set Angle (PASA),Distal Articular Set Angle(DASA), and the metatarsophalangeal angle of the first ray (lateral projection).

Materials and Methods: The chosen study design is an experimental, controlled, non-randomized, longitudinal, analytical, and prospective study. Subjects meeting the selection criteria will be non-randomly assigned to two different groups: the "Minimally Invasive Surgery Group with Zig-zag EHL Tenotomy" and the "Minimally Invasive Surgery Group without Zig-zag EHL Tenotomy." After surgery, a follow-up with radiological control will be performed, where post-surgical angles will be measured and plantar pressures will be evaluated.

Results: The investigators expect to achieve effective and safe lengthening of the long hallux extensor in all patients with HAV and hyperextension of the first toe.

Conclusions: The study results will indicate that zig-zag tenotomy of the long hallux extensor is a safe, effective, and rapid technique.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the metatarsophalangeal joint of the big toe caused by HAV.
* Moderate and severe Hallux Abductus Valgus.
* Incorrect metatarsal shape of the 2nd, 3rd and 4th rays due to HAV.
* Be between 20 and 90 years old.
* Patients with no osteoarthritis.

Exclusion Criteria:

* Patients who have previously undergone surgery for Hallux Abductus Valgus.
* Pregnant patients.
* Patients with coagulopathies, diabetes or risk disease (ASA lll, ASA lV).
* Patients with high-risk pharmacological treatments.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this project is men and women between 20 and 90 years old with hallux abductus valgus and the first toe in hyperextension on one or both feet. The subjects in the sample will be patients undergoing surgery in private clinics who come for consultation at the time of the study. The method to select the sample is non-probabilistic due to the inclusion of volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Radiographic | Pre-surgery, 2 months, 6months
  Flat Panel is a direct digitization radiography system that provides us with the image in two seconds. The investigators will perform dorso-plantar and lateral oblique radiographs of the patients' feet.

SECONDARY OUTCOMES:
Pressure platform | Pre-surgery, 2 months, 6months
  It is a tool that allows us to know the distribution of pressures on the sole of the foot, both statically and dynamically. It offers a range of colors in the patient's footprint according to the baropressure captured. It will help us determine the change in pre-surgical and post-surgical plantar pressures.
American Orthopedic Foot and Ankle Society | Pre-surgery, 2 months, 6months
  This questionnaire incorporates subjective and objective factors that are scored using a numerical scale and describe variables of function, alignment and pain. The score ranges from 0 to 100 depending on the degree of limitation of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Ferrer-Torregrosa, Dr., Study Director — Fundación Universidad Católica de Valencia San Vicente Mártir
Locations (1):
- Levante Salud, Ondara, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marijuschkin I, Souza ML, Diaz JLG, Carvalho P. Percutaneous Hallux Valgus: An Algorithm for the Surgical Treatment. Rev Bras Ortop (Sao Paulo). 2021 Aug;56(4):504-512. doi: 10.1055/s-0040-1721367. Epub 2021 Aug 30. PMID 34483396
- [Background] Restuccia G, Lippi A, Sacchetti F, Citarelli C, Casella F, Benifei M. Percutaneous Hallux Valgus Correction: Modified Reverdin-Isham Osteotomy, Preliminary Results. Surg Technol Int. 2017 Dec 22;31:263-266. PMID 29310149
- [Background] Bauer T, Biau D, Lortat-Jacob A, Hardy P. Percutaneous hallux valgus correction using the Reverdin-Isham osteotomy. Orthop Traumatol Surg Res. 2010 Jun;96(4):407-16. doi: 10.1016/j.otsr.2010.01.007. Epub 2010 May 20. PMID 20488776
- [Background] Botezatu I, Marinescu R, Laptoiu D. Minimally invasive-percutaneous surgery - recent developments of the foot surgery techniques. J Med Life. 2015;8 Spec Issue(Spec Issue):87-93. PMID 26361518
- [Background] Maffulli N, Longo UG, Marinozzi A, Denaro V. Hallux valgus: effectiveness and safety of minimally invasive surgery. A systematic review. Br Med Bull. 2011;97:149-67. doi: 10.1093/bmb/ldq027. Epub 2010 Aug 14. PMID 20710024
- [Background] Biz C, Fosser M, Dalmau-Pastor M, Corradin M, Roda MG, Aldegheri R, Ruggieri P. Functional and radiographic outcomes of hallux valgus correction by mini-invasive surgery with Reverdin-Isham and Akin percutaneous osteotomies: a longitudinal prospective study with a 48-month follow-up. J Orthop Surg Res. 2016 Dec 5;11(1):157. doi: 10.1186/s13018-016-0491-x. PMID 27919259
- [Background] Lu J, Zhao H, Liang X, Ma Q. Comparison of Minimally Invasive and Traditionally Open Surgeries in Correction of Hallux Valgus: A Meta-Analysis. J Foot Ankle Surg. 2020 Jul-Aug;59(4):801-806. doi: 10.1053/j.jfas.2019.03.021. PMID 32600562
- [Background] Bia A, Guerra-Pinto F, Pereira BS, Corte-Real N, Oliva XM. Percutaneous Osteotomies in Hallux Valgus: A Systematic Review. J Foot Ankle Surg. 2018 Jan-Feb;57(1):123-130. doi: 10.1053/j.jfas.2017.06.027. Epub 2017 Sep 1. PMID 28870735
- [Derived] Sanchis-Soria V, Ferrer-Torregrosa J, Marti-Martinez LM, Carratala-Villarroya G, Vicente-Mampel J, Lorca-Gutierrez R. Multimodal evaluation of partial zig-zag tenotomy of the extensor hallucis longus in minimally invasive hallux valgus surgery: a randomized trial. J Orthop Surg Res. 2025 Nov 28;21(1):3. doi: 10.1186/s13018-025-06456-x. PMID 41316331